CLINICAL TRIAL: NCT04912934
Title: The Relationship Between Coronavirus Anxiety Level and Emotional Eating in Individuals With Metabolic Syndrome
Brief Title: The Relationship Between COVID-19 Anxiety Level and Emotional Eating in Individuals With Metabolic Syndrome
Acronym: COVID-19
Status: Completed | Type: Observational
Sponsor: Ordu University (Other)
Responsible Party: Principal Investigator, Dilekkucu Kalemdar, Associate Professor, Ordu University
Other Study IDs: KAEK-228
Record Dates: First submitted 2021-05-30; First posted 2021-06-03 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2021-06

CONDITIONS: Metabolic Syndrome; Emotional Eating; COVID-19
Keywords: Metabolic Syndrome; COVID-19; Eating
MeSH Terms: conditions — Metabolic Syndrome; Emotional Eating; COVID-19 | interventions — Glucose; oxidized low density lipoprotein; Cholesterol; Triglycerides; Insulin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — glucose, HDL, LDL, total cholesterol, triglycerides, CRP, HbA1c, insulin, HOMA-IR
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MetS diagnosis: The research included individuals aged 18 years and older, who were not pregnant or breastfeeding, without any psychological disorder diagnosed by psychiatry, without diagnosis of COVID-19 and not using any psychiatric medications. The MetS group for the research included individuals with metabolic syndrome diagnosis according to IDF-2005 diagnostic criteria.
  Interventions: Procedure: A survey form was applied to individuals included in the study face-to-face.
- non-MetS: The research included individuals aged 18 years and older, who were not pregnant or breastfeeding, without any psychological disorder diagnosed by psychiatry, without diagnosis of COVID-19 and not using any psychiatric medications. The non MetS group in the research included healthy individuals not using any psychiatric medications, without any chronic disorder, and with similar BMI to the individuals in the subject group.
  Interventions: Procedure: A survey form was applied to individuals included in the study face-to-face.

INTERVENTIONS:
Procedure: A survey form was applied to individuals included in the study face-to-face. — This study was completed with a descriptive, cross-sectional and relational screening model
  Other Names: This survey form; Biochemical findings (glucose, HDL, LDL, total cholesterol, triglycerides, CRP, HbA1c, insulin, HOMA-IR).; Blood pressure was measured and recorded.; The coronavirus anxiety scale (CAS) and emotional eating scale (EES) were applied.

SUMMARY:
The aim was to determine the coronavirus anxiety levels and emotional eating status of cases with diagnosis of MetS according to diagnostic criteria published by the International Diabetic Federation (IDF) in 2005 and healthy individuals with similar BMI to MetS subjects.

DETAILED DESCRIPTION:
The aim was to determine the coronavirus anxiety levels and emotional eating status of cases with diagnosis of MetS according to diagnostic criteria published by the International Diabetic Federation (IDF) in 2005 and healthy individuals with similar BMI to MetS subjects. This study was completed with the descriptive, cross-sectional and relational screening model. The full sampling method was used in the study. The study was completed with 105 individuals with metabolic syndrome attending the diet clinic and 109 healthy individuals without MetS diagnosis also attending the diet clinic. Collection of data used anthropometric measurements and biochemical findings, blood pressure and a survey form, the Coronavirus Anxiety Scale (CAS) and Emotional Eating Scale (EES).

ELIGIBILITY:
Inclusion Criteria:

* The research included individuals aged 18 years and older, who were not pregnant or breastfeeding, without any psychological disorder diagnosed by psychiatry, without diagnosis of COVID-19 and not using any psychiatric medications. The MetS group for the research included individuals with metabolic syndrome diagnosis according to IDF-2005 diagnostic criteria. The non MetS group in the research included healthy individuals not using any psychiatric medications, without any chronic disorder, and with similar BMI to the individuals in the subject group.

Exclusion Criteria:

* The research included individuals aged 18 years and older, who were pregnant or breastfeeding, with psychological disorder diagnosed by psychiatry, with diagnosis of COVID-19 and using psychiatric medications.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Power analysis was performed using the G*Power (v3.1.9) program to determine the number of samples. According to Jacob Cohen's effect size coefficients, it was calculated that there should be at least 105 people in the groups for α=0.05 and 1-β=0.95 (95% power) levels, assuming that the evaluations between the two independent groups would have a medium effect size (d=0.5).
Sampling Method: Non-Probability Sample
Enrollment: 214 (Actual)
Dates: Start 2020-06-20 (Actual); Primary Completion 2020-11-20 (Actual); Study Completion 2020-12-12 (Actual)

PRIMARY OUTCOMES:
Coronavirus anxiety scale (CAS) | 5 month
  Total points of ≥9 on the scale shows dysfunctional anxiety related to coronavirus.
Emotional eating scale (EES) | 5 month.
  High points on the scale show high levels of emotional eating behavior.

SECONDARY OUTCOMES:
BMI (Body Mass Index) | 5 month.
  kg/m^2
Glucose | 5 month.
  mg/dL
Blood pressure | 5 month.
  Systolic and diastolic blood pressure
HDL | 5 month.
  mg/dL
LDL | 5 month.
  mg/dL
triglycerides | 5 month.
  mg/dL
HbA1c | 5 month.
  HbA1c (%)
insulin | 5 month.
  ng/ml
HOMA-IR | 5 month.
  index
total cholesterol | Through study completion, an average of 5 month.
  mg/dL
CRP | 5 month.
  mg/dL

CONTACTS AND LOCATIONS:
Overall Officials: Dilek Küçük Alemdar, Study Director — Ordu University
Locations (1):
- Dilek alemdar, Ordu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang J, Zhang Y, Huo S, Ma Y, Ke Y, Wang P, Zhao A. Emotional Eating in Pregnant Women during the COVID-19 Pandemic and Its Association with Dietary Intake and Gestational Weight Gain. Nutrients. 2020 Jul 28;12(8):2250. doi: 10.3390/nu12082250. PMID 32731389